CLINICAL TRIAL: NCT04870073
Title: Retrograde Autologous Priming for Preserving Hemoglobin Peri-operatively With or Without Mannitol: A Pilot Study
Brief Title: Retrograde Autologous Priming and Mannitol for Reducing Hemodilution in Cardiac Surgery
Acronym: RAPPER-MAN
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Financial support could not be obtained for the study
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Andre Lamy, Cardiac Surgeon, Hamilton Health Sciences Corporation
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RAPPER-MAN_2021
Record Dates: First submitted 2021-04-20; First posted 2021-05-03 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Hemodilution; Coronary Artery Disease; Fluid Overload
Keywords: retrograde autologous priming; mannitol; cardiopulmonary bypass; cardiac surgery; hemodilution
MeSH Terms: conditions — Coronary Artery Disease; Edema | interventions — Mannitol

STUDY DESIGN:
Intervention Model Description: single-centre, single blinded, 2x2 factorial, cluster randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Retrograde autologous priming + mannitol (Experimental): Priming solution (≥600 mL) will be removed from the extracorporeal circuit within 10 minutes before the initiation of cardiopulmonary bypass. Priming solution may be removed from 3 locations within the extracorporeal circuit (i.e. arterial, venous and cardioplegia lines) as determined by the perfusionist team. In addition, mannitol will be added as a bolus (0.3 g/kg) to the venous reservoir of the cardiopulmonary bypass machine within 5 min before the start of cardiopulmonary bypass.
  Interventions: Procedure: Retrograde autologous priming; Drug: Mannitol
- Retrograde autologous priming alone (Experimental): Priming solution (≥600 mL) will be removed from the extracorporeal circuit within 10 minutes before the initiation of cardiopulmonary bypass. Priming solution may be removed from 3 locations within the extracorporeal circuit (i.e. arterial, venous and cardioplegia lines) as determined by the perfusionist team.
  Interventions: Procedure: Retrograde autologous priming
- Conventional priming + mannitol (Experimental): Participants will receive conventional priming. In addition, mannitol will be added as a bolus (0.3 g/kg) to the venous reservoir of the cardiopulmonary bypass machine within 5 min before the start of cardiopulmonary bypass.
  Interventions: Drug: Mannitol; Procedure: Conventional Priming
- Conventional priming alone (Active Comparator): Participants will receive conventional priming alone.
  Interventions: Procedure: Conventional Priming

INTERVENTIONS:
Procedure: Retrograde autologous priming — Priming solution (≥600 mL) will be removed from the extracorporeal circuit within 10 minutes before the initiation of cardiopulmonary bypass. Priming solution may be removed from 3 locations within the extracorporeal circuit (i.e. arterial, venous and cardioplegia lines) as determined by the perfusionist team.
  Other Names: RAP
  Arms: Retrograde autologous priming + mannitol; Retrograde autologous priming alone
Drug: Mannitol — Mannitol will be added as a bolus (0.3 g/kg) to the venous reservoir of the cardiopulmonary bypass machine within 5 min before the start of cardiopulmonary bypass.
  Arms: Conventional priming + mannitol; Retrograde autologous priming + mannitol
Procedure: Conventional Priming — The conventional priming procedure will be used in the standardized cardiopulmonary machine used at the Hamilton General Hospital.
  Arms: Conventional priming + mannitol; Conventional priming alone

SUMMARY:
Hemodilution reduces concentrations of blood constituents: concentration of hemoglobin, red blood cells (hematocrit), physiological ions and coagulation factors that can contribute to impaired hemostasis and increasing the risk of perioperative blood transfusions. This pilot study will assess the feasibility of a large RCT to evaluate 2 techniques for reducing hemodilution during cardiac surgery: 1) retrograde autologous priming and 2) intraoperative mannitol. The aim of this pilot trial is to demonstrate feasibility of a larger trial to evaluate whether retrograde autologous priming and/or mannitol are superior to conventional priming alone.

DETAILED DESCRIPTION:
The use of large volumes of artificial priming fluids is still very high in cardiac surgery for routine CABG surgery with cardiopulmonary bypass. The resulting hemodilution is deleterious for patients and often requires counter measures to maintain fluid balance during and after surgery. Retrograde autologous priming and mannitol are simple low-cost solutions to the problem of hemodilution but their effectiveness, either alone or in combination, is unclear due to a lack of high-quality evidence. RAPPER-MAN is a single-centre 2x2 factorial cluster randomized trial. Participants will be randomly assigned (1:1:1:1 ratio) to the intervention groups: 1) Retrograde autologous priming (≥600 mL) + mannitol (0.3 g/kg bolus), 2) Retrograde autologous priming (≥600 mL) alone, 3) Conventional priming + mannitol (0.3 g/kg bolus), and 4) Conventional priming alone. The primary outcome is the change in hemoglobin concentration during cardiopulmonary bypass. Retrograde autologous priming will be performed within 10 minutes before, and mannitol will be added to the venous reservoir of the CPB machine within 5 minutes before, the start of cardiopulmonary bypass. The results of the larger trial are expected to have broad implications for fluid management in cardiac surgery in Canada.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age.
2. Undergoing a first-time cardiac surgical procedure (i.e. isolated CABG, isolated single cardiac valve surgery or a combination of both or isolated ascending aorta replacement) with the use of cardiopulmonary bypass (CPB) and median sternotomy.

Exclusion Criteria:

1. Left ventricle ejection fraction <25%
2. Emergency surgery
3. History of bleeding disorder
4. Inherited thromboembolic or infective endocarditis (active)
5. Previous cardiac surgery
6. Severe renal impairment (serum creatinine >250 μmol/L)
7. Hemoglobin <80 g/L
8. Thrombocytopenia (<50,000 platelets per μL)
9. Expected circulatory arrest
10. Body weight ≤50 kg
11. Allergy to mannitol
12. Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2022-09-21 (Actual)

PRIMARY OUTCOMES:
Feasibility Outcomes | Start to end of study recruitment, which is anticipated to take 20 weeks
  Feasibility will be established in the pilot phase if all the following criteria are met:
  1. Average recruitment rate of 7 patients per week.
  2. Complete Hb data before and after cardiopulmonary bypass in 90% of patients.
  3. Compliance of the research team members, OR staff and ward medical staff with the protocol of 90%.
Change in hemoglobin concentration during cardiopulmonary bypass | Start to end of cardiopulmonary bypass
  Change in arterial hemoglobin concentration during cardiopulmonary bypass

SECONDARY OUTCOMES:
Change in hemoglobin concentration after cardiopulmonary bypass | Start of cardiopulmonary bypass to hospital discharge or 5 days maximum (whichever occurs first)
  Change in arterial hemoglobin concentration from baseline to discharge

OTHER OUTCOMES:
Blood transfusion | Start of surgery to hospital discharge or 5 days maximum (whichever occurs first)
  Proportion of patients experiencing red blood cell transfusion
Change in oxygen consumption during cardiopulmonary bypass | Start to end of cardiopulmonary bypass
  Change in oxygen consumption during cardiopulmonary bypass
Autologous prime volume | Within 10 minutes before cardiopulmonary bypass
  Total prime volume removed from the extracorporeal circuit during the retrograde autologous priming procedure
Hyponatremia | Before and 24 hours after surgery
  Sodium concentration of less than 135 mmol/L (135 mEq/L)
Diuresis | Within 24 hours of surgery
  Total volume of urine within 24 hours of surgery
Hemofiltration use | During cardiopulmonary bypass
  Proportion of patients undergoing hemofiltration
Fluid balance | Daily in ICU from admission to hospital discharge or 5 days maximum (whichever occurs first)
  Net fluid balance (intake minus output) calculated using a cumulative fluid chart
Acute kidney injury | Start of surgery to hospital discharge or 5 days maximum (whichever occurs first)
  Acute kidney injury as measured by peak postoperative creatinine and KDIGO
Length of hospital stay | Time from admission to hospital discharge or 5 days maximum (whichever occurs first)
  Length of hospital stay (days)
Major adverse cardiovascular events | Start of surgery to hospital discharge or 5 days maximum (whichever occurs first)
  Composite outcome of cardiovascular death, non-fatal myocardial infarction or stroke

CONTACTS AND LOCATIONS:
Overall Officials: Andre Lamy, MD, Principal Investigator — Hamilton Health Sciences Corporation
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hensley NB, Gyi R, Zorrilla-Vaca A, Choi CW, Lawton JS, Brown CH 4th, Frank SM, Grant MC, Cho BC. Retrograde Autologous Priming in Cardiac Surgery: Results From a Systematic Review and Meta-analysis. Anesth Analg. 2021 Jan;132(1):100-107. doi: 10.1213/ANE.0000000000005151. PMID 32947294
- [Background] Ljunggren M, Skold A, Dardashti A, Hyllen S. The use of mannitol in cardiopulmonary bypass prime solution-Prospective randomized double-blind clinical trial. Acta Anaesthesiol Scand. 2019 Nov;63(10):1298-1305. doi: 10.1111/aas.13445. Epub 2019 Jul 29. PMID 31287556
- [Background] Task Force on Patient Blood Management for Adult Cardiac Surgery of the European Association for Cardio-Thoracic Surgery (EACTS) and the European Association of Cardiothoracic Anaesthesiology (EACTA); Boer C, Meesters MI, Milojevic M, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Pagano D. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. J Cardiothorac Vasc Anesth. 2018 Feb;32(1):88-120. doi: 10.1053/j.jvca.2017.06.026. Epub 2017 Sep 30. No abstract available. PMID 29029990
- [Background] Trapp C, Schiller W, Mellert F, Halbe M, Lorenzen H, Welz A, Probst C. Retrograde Autologous Priming as a Safe and Easy Method to Reduce Hemodilution and Transfusion Requirements during Cardiac Surgery. Thorac Cardiovasc Surg. 2015 Oct;63(7):628-34. doi: 10.1055/s-0035-1548731. Epub 2015 Mar 24. PMID 25803120